CLINICAL TRIAL: NCT00422825
Title: A Phase I, Open-label, Randomized, Crossover Study to Investigate the Effect of Food on the Bioavailability of a Single 800 mg Imatinib Dose in a Modified Release Formulation (MR2) and Compare the Bioavailability Between MR2 and Imatinib 400 mg Twice Daily Immediate Release Tablet (IR) in Healthy Subjects
Brief Title: Effect of Food on Bioavailability of a Modified Release Formulation of Imatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571O2102
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Food effect; bioavailability; pharmacokinetic; imatinib; STI571; modified release formulation of STI571; CML; Chronic Myeloid Leukemia; Philadelphia Chromosome
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imatinib 800mg (Experimental)
  Interventions: Drug: imatinib
- Imatinib 400mg (Active Comparator)
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: imatinib

SUMMARY:
This is a single center, four-treatment, four period, crossover study to evaluate the effect of food on the relative bioavailability of a single dose of imatinib (STI571) given as a 800 mg modified release tablet, MR2 compared to twice-daily doses of 400 mg film-coated imatinib tablets. There will be a 10 day wash out phase between treatments and a 1 week safety period at the end of the study. Each participant will receive all four treatments

ELIGIBILITY:
Inclusion criteria

* Healthy male or female subjects (postmenopausal women)
* Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion criteria

* Smokers
* Subjects using any prescription drug or over-the-counter (OTC) medication (including herbal and alternative medication) within 2 weeks prior to dosing.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* A past medical history or presence of clinically significant ECG abnormalities including:
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* History of medications pre-disposing the subjects for GI bleedings/cerebral hemorrhage.
* Women taking any biphosphonates (Fosomax like drugs)
* History of being immunocompromised, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* Females nursing infants. Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Assess the effect of food on bioavailability and pharmacokinetics of modified and immediate release formulations of imatinib

SECONDARY OUTCOMES:
To compare safety and tolerability of 800 mg modified release formulation with or without food.
To compare the relative bioavailability of a single dose 800 mg modified release formulation (with a low fat breakfast) with the marketed 400 mg immediate release tablet administered (with a low fat breakfast) twice daily

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis